CLINICAL TRIAL: NCT02640469
Title: Efficacy of the Use of Alcohol-bases Solutions Versus Chlorhexidine With or Without Water for Hand Sanitation Prior to Surgical Procedure
Brief Title: Alcohol Versus Chlorhexidine With and Without Water
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 14-00496
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Infection
Keywords: chlorhexidine; sterility; sterile hands
MeSH Terms: conditions — Infections; Infertility | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine with water rinse (Active Comparator): This is a traditional method of disinfection used at NYU Hospital for Joint Disease. Following disinfection protocol, each subject will have hand cultured three times using a cotton swab culture and sent to microbiology for processing.
  Interventions: Other: Chlorhexidine with water rinse
- Chlorhexidine without water rinse (Experimental): This is an experimental method of disinfection. Following disinfection protocol, each subject will have hand cultured three times using a cotton swab culture and sent to microbiology for processing.
  Interventions: Other: Chlorhexidine without water rinse
- Chlorhexidine + sterillium hand rub (Active Comparator): This is a standard method of disinfection used at NYU Hospital for Joint Disease. Following disinfection protocol, each subject will have hand cultured three times using a cotton swab culture and sent to microbiology for processing.
  Interventions: Other: Chlorhexidine + sterillium hand rub

INTERVENTIONS:
Other: Chlorhexidine with water rinse — This procedure will be followed for both the right and left hands and arms:
  scrub each side of finger, in between fingers and back and front of hands for 2 minutes, followed by scrubbing of arms, keeping hands higher than arms at all times, wash each side of the arms from wrist to elbow for 1 minute
  Arms: Chlorhexidine with water rinse
Other: Chlorhexidine without water rinse — Scrub each side of finger, in between fingers and back and front of hands for 2 minutes, proceed to scrub the arms, keeping the hand higher than the arm at all times, wash each side of the arms from wrist to elbow for 1 minute, and repeat the process on the other arm.
  Arms: Chlorhexidine without water rinse
Other: Chlorhexidine + sterillium hand rub — Scrub each side of finger, in between fingers and back and front of hands for 2 minutes, Scrub each side of finger, in between fingers and back and front of hands for 2 minutes, proceed to scrub the arms, keeping the hand higher than the arm at all times, wash each side of the arms from wrist to elbow for 1 minute, and repeat the process on the other arm. Rinse hands and arms by passing through water in one direction, dry hands, and rub 5 mL of alcohol into the palm of the hands, forearms and elbows. Ensure that the whole skin area on both arms is covered.
  Arms: Chlorhexidine + sterillium hand rub

SUMMARY:
Currently at NYU institutions, providine-iodine and chlorhexidine medicated soaps are available as hand disinfection options. The purpose of this study is to determine the relative efficacy of traditional hand scrubs with chlorhexidine with or without rinsing with water after scrubbing is complete versus dry hand rubs with alcohol.

DETAILED DESCRIPTION:
No current recommendations exist advocating the use of Providine-iodine or Chlorhexidine. Providine-iodine is safe and effective at reducing skin colonization with gram positive and negative bacteria, mycobacterium tuberculosis, fungi and viruses. Chlorhexidine similarly disrupts cellular membranes. It is bacteriocidal and bacteriostatic and has immediate and more lasting effect than iodine because it can bind to the stratum corneum of the skin and is effective against gram positive and negative organisms, lipophilic viruses and yeasts.

All subjects who are employees of the NYU Hospital for Joint Diseases and have experience with surgical hand disinfection will be asked to enroll. Subjects will be randomized into one of three study arms using an online randomizer: (1) the standard chlorhexidine with water rinse, (2) chlorhexidine without water rinse(experimental), and (3) standard chlorhexidine followed by sterillium hand rub. After hand disinfection protocol has been completed, each subject will have each hand cultured three times using a cotton swab culture stick and sent to the microbiology lab for processing

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic resident or surgical employee of NY U
* Over 21 years of age
* Procedural knowledge of correct aseptic scrub technique

Exclusion Criteria:

* No surgical experience
* Under 21 years of age
* Refusal to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Number of positive cultures in each group | 1 day
  Evaluated using a Students T-test and analysis of variance (ANOVA).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Liporace, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University Hospital for Joint Disease, New York, New York, United States